CLINICAL TRIAL: NCT02996760
Title: Influence Instillation Plasma Rich in Growth Factors in Endometrial Cavity
Brief Title: Influence Instillation Plasma Rich in Growth Factors in Endometrial Cavity Endometrial Development in Assisted Reproduction.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulty in recruiting
Sponsor: IVI Bilbao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1404-BIO-019-MF
Record Dates: First submitted 2016-12-02; First posted 2016-12-19 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Endometrial Development
MeSH Terms: interventions — Platelet-Derived Growth Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometrium with less than 5mm (Experimental): Women receiving cycle of oocytes outside or embryos (own / others), in the treatment of substituted cycle type.
  Less than 5mm despite 10 days with standard doses of estrogen
  Interventions: Drug: Growth Factor, Platelet-Derived
- Endometrium with more than 5mm (No Intervention): Women receiving cycle of oocytes outside or embryos (own / others), in the treatment of substituted cycle type.
  More than 5mm despite 10 days with standard doses of estrogen

INTERVENTIONS:
Drug: Growth Factor, Platelet-Derived — 0,5 mL, vaginal use , 3 dose number
  Arms: Endometrium with less than 5mm

SUMMARY:
Women in assisted reproduction treatment they receive own or donated embryos and presenting an endometrial development less than 5 mm despite having received treatment with estrogen therapy knowing the clinical value of using the PRGF-Endoret therapy and endometrial level applications to improve endometrial thickness endometrial preparations for embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Women receiving cycle of oocytes outside or embryos (own / others), in the treatment of substituted cycle type.
* Less than 5mm despite 10 days with standard doses of estrogen therapy (6mg / 24h) Endometrio

Exclusion Criteria:

* History of pelvic inflammatory disease
* Risk of infection

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the growth of endometrial thickness | During ovarian stimulation protocol 8-12 days
  The endometrial thickness will be measured by vaginal ultrasound. Endometrium less than 5 mm will be treated

SECONDARY OUTCOMES:
Analyze the impact of using platelet plasma on rates of implantation and pregnancy. | During ovarian stimulation protocol 8-12 days
  The biochemical determination of the hormone ßhcg will be performed 12 days after embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Bilbao, Leioa, Vizcaya, Spain